CLINICAL TRIAL: NCT06230484
Title: A Prospective Clinical Trial on the Outcomes of Invisalign First Palatal Expander
Brief Title: IFPE (Invisalign First Palatal Expander)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Bingshuang Zou, Principal Investigator, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H23-00231
Record Dates: First submitted 2024-01-07; First posted 2024-01-30 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Narrow Maxilla

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- IFPE patients (Active Comparator): patients receiving IFPE treatment
  Interventions: Device: Invisalign first palatal expander
- (control group): RME patients (Active Comparator): patients receiving conventional rapid maxillary expansion treatment
  Interventions: Device: Conventional rapid maxillary expansion

INTERVENTIONS:
Device: Invisalign first palatal expander — Most recently, a new design of a removable expander by Align was brought to our attention. In this prospective clinical study, the investigators will compare the patient-reported treatment outcomes and the dental-skeletal treatment effects on palatal dimensions. With this study, the investigators will have a better understanding of this newly developed appliance and its application in early orthodontic treatment.
  Arms: IFPE patients
Device: Conventional rapid maxillary expansion — Malocclusions with narrow upper arches are usually treated in the mixed dentition with a traditional bonded maxillary expander.
  Arms: (control group): RME patients

SUMMARY:
Malocclusions with narrow upper arches are usually treated in the mixed dentition with a traditional bonded maxillary expander. Most recently, a new design of a removable expander by Align was brought to our attention. In this prospective clinical study, the investigators will compare the patient-reported treatment outcomes and the dental-skeletal treatment effects on palatal dimensions. With this study, the investigators will have a better understanding of this newly developed appliance and its application in early orthodontic treatment.

DETAILED DESCRIPTION:
Purpose:

This prospective study is aimed to investigate the patient-reported treatment outcomes and the dental-skeletal treatment effects on palatal dimensions and to compare them with those of traditional maxillary expansion.

Hypothesis:

The null hypothesis will be:

* 1: There are no differences in the inter-canine, inter-molar width, and molar inclination between IFPE and RME groups.
* 2: There are no differences in the arch width, length, size and shape, palatal surface area and volume, plaque index, and white spot lesion formation between IFPE and RME groups.
* 3: There are no differences in patients' experience of perceived pain intensity and discomfort during the first two weeks of treatment between IFPE and RME groups.

Justification:

The Invisalign First System (IFS) has been used in transverse arch development but with less skeletal effects in growing subjects. A new appliance, Invisalign First palatal expander (IFPE), designed to rapidly expand the maxillary arch with a daily change protocol has been introduced. This prospective clinical trial will compare the efficacy and efficiency between IFPE and conventional rapid maxillary expansion (RME) for maxillary arch expansion in mixed dentition. Patient-reported treatment outcomes in terms of quality of life during the treatment will also be investigated.

Objectives:

The broad, long-term objective of the project is to evaluate the efficacy and efficiency of IFPE and compare the treatment outcomes with those of subjects treated with conventional RME.

The specific aim of this research project is to compare the primary (the inter-molar width, molar inclination, the arch width, length, size and shape, palatal surface area and volume) and secondary (plaque index, and white spot lesion formation, difficulties with speech and eating) outcomes between IFPE and conventional RME for maxillary arch expansion in mixed dentition. With the results of this prospective clinical trial, orthodontists will gain knowledge of the efficacy and efficiency of IFEP compared with traditional RME and make their own decisions with the evidence to be provided by this study.

Research Protocol:

Research Design:

A power calculation based on the previous study by Lione et al.12 indicated a sample of 50 patients in each group to estimate inter-first molar width with a minimum difference of 1mm and a standard deviation (SD) of 3mm, with a power of 80%.

This project will be a multi-centre, prospective clinical trial with two parallel arms. The study protocol will be registered on CliniclTrials.gov. Ethical approval will be obtained from the Institute Research Board of the University of British Columbia before trial commencement and informed consent will be required from each subject before entering the study.

The recruitment will occur at two private orthodontic offices: one is an Invisalign diamond provider's office, and the other is a pediatric dentist and orthodontist group office. All the patients who meet the eligibility criteria will be treated with IFPE in the first office. While patients recruited from the second office under the same inclusion criteria will be treated with conventional Hyrax-type RME. The eligibility criteria will include patients of both sexes from 6 - 12 years of age, in mixed dentition with maxillary first molars completely erupted, and transverse maxillary deficiency. In particular, the presence of unilateral or bilateral crossbite, or intermolar width (as measured where the palatal groove meets the gingival margin of the first molar) of 33 mm or less). Exclusion criteria will include the following: multiple and/or advanced caries, missing teeth due to aplasia, trauma, or deep caries, supernumerary teeth, congenital craniofacial malformations or congenital or acquired systematic disease, and previous orthodontic treatment.

For each group, 50 consecutively recruited patients will be treated with IFPE and RME, respectively. For the IFPE group, patients will be treated with IFPE with no other auxiliaries and no enamel interproximal reduction (IPR) will be planned during treatment. Patients will be instructed to wear the expander 20-22 hours/day with a daily change protocol until the maxillary lingual cusps are in contact with the mandibular buccal cusps, followed by passive retention for 6 months. In the RME group, a two-banded Hyrax-type expander with one-quarter turn (0.25mm) every day will be performed until the maxillary lingual cusps are in contact with the mandibular buccal cusps, followed by a passive retention of 6 months. Orthodontic appointments will be scheduled weekly at first, then moved to monthly.

Digital casts before (T1) and after expansion (T2) will be collected and inter-canine width, inter-molar width, molar inclination, palatal width, surface area, and volume will be measured by using Rhino3D v5.0 software (Robert McNeel and Associates, Seattle, Wash). The buccal surfaces of the maxillary molars will be assessed for non-cavitated carious lesions (white spot lesions) using the International Caries Detection and Assessment System (ICDAS) index. The plaque index was assessed using color-based plaque staining. Questionnaires will be given to the patients to fill out on days 1, 7 and 14 regarding level of pain and discomfort, difficulty with speech and eating, interference with daily activities and functional jaw impairment.

Statistical analysis:

SPSS software (version 27.0, IBM Corp. Armonk, NY) will be used for the statistical analyses. Measurements for 10 randomly selected models will be repeated 1 week apart to assess intra-examiner agreement. Intra-class correlation coefficients and Bland-Altman plots will be used to test the intra-examiner agreement. All measurements will be assessed for normality using the Shapiro-Wilks test. Descriptive statistics in the form of median and interquartile ranges (IQR, Q3-Q1) will be reported when the parameters did not show a normal distribution. Changes between T1 and T2 in each group will be analyzed with paired t-test for normal data and Wilcoxon signed-rank test for non-normal data. Intergroup comparison will be evaluated with t-tests or Mann-Whitney U-tests with Bonferroni correction. The significant level was set as P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients in mixed dentition with 6 present on both Right and Left in the upper arch
* Patients with transverse maxillary deficiency (presence of unilateral or bilateral crossbite, or intermolar width (as measured where the palatal groove meets the gingival margin of the first molar) of 33 mm or less)

Exclusion Criteria:

* multiple and/or advanced caries,
* missing teeth due to aplasia, trauma, or deep caries,
* supernumerary teeth,
* congenital craniofacial malformations or congenital or acquired systematic disease,
* previous orthodontic treatment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
inter-canine, inter-molar, and palatal width | one year
  measured by using Rhino3D v5.0 software in millimeters
Qualitative measurements from questionnaire- level of pain and discomfort | one year
  VAS = visual analogue scale, ranges from minimum score 0% (extremely uncomfortable) to 100% (very comfortable). Higher score is good (comfortable).
molar inclination | one year
  measured by using Rhino3D v5.0 software in degrees
surface area | one year
  measured by using Rhino3D v5.0 software in millimeters squared
volume | one year
  measured by using Rhino3D v5.0 software in millimeters cubed
noncavitated carious lesions | one year
  The buccal surfaces of the maxillary molars will be assessed for noncavitated carious lesions (white spot lesions) using the International Caries Detection and Assessment System (ICDAS) index. The higher the score the worse condition:
  0 Sound
  1. First visual change in enamel (seen only after prolonged air drying or restricted to the confines of a pit or fissure)
  2. Distinct visual change in enamel
  3. Localized enamel breakdown (without clinical visual signs of dentinal involvement)
  4. Underlying dark shadow from dentin
  5. Distinct cavity with visible dentin
  6. Extensive distinct cavity with visible dentin
Plaque | one year
  Plaque index was assessed using color-based plaque staining. 0 - no visible plaque, 1-plaque visible only by scraping on the denture base with a blunt instrument, 2-moderate accumulation of visible plaque, and 3-abundance of plaque. By summing up the scores from the five areas, the plaque was recorded on a scale from 0 to 15 points.

IPD SHARING:
Plan to Share IPD: No